CLINICAL TRIAL: NCT06839846
Title: Survey of Different Modes of Weaning in Pediatric Population
Acronym: DIVPED
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: DIVPED
Record Dates: First submitted 2024-12-01; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-10

CONDITIONS: Weaning
Keywords: weaning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parents: the survey will be proposed to adult parents of children aged 4-18 months by means of a specific questionnaire dedicated to them.
- Pediatrician: another specific questionnaire intended for the Pediatrician will be proposed to PLSs who give their willingness.

SUMMARY:
Infant weaning refers to the transition from a diet based on the exclusive intake of milk (mother's milk or formula) to a diversified diet that is complete with all the nutrients necessary for proper infant development. For this purpose, a diet supplementary to milk, which is gradually reduced, is undertaken in order to gradually acquire the dietary pattern followed by the family.

There are different types of weaning, which vary according to traditions, ethnicity and scientific currents. These include traditional weaning and on-demand self-weaning. The former consists of weaning with specific infant foods (example: freeze-dried, homogenized, vegetable broth, creams..) offered at set doses, quantities, and times. On the other hand, 'autodivezzamento on demand is a mode of weaning entrusted to the child's request, leaving the child to choose quantities and types of food, even prepared at home, during family meals. The aim of our study is to establish the prevalence of different modes of weaning and the perception of advantages and disadvantages related to them by parents and Free Choice Pediatricians by means of two different dedicated questionnaires. The study also aims to assess possible risks resulting from the transition to complementary feeding, for example, errors in feeding or inhalation of foreign bodies.

DETAILED DESCRIPTION:
Infant weaning refers to the transition from a diet based solely on milk (breast milk or formula) to a diversified and complete diet, given by the presence of all foods introduced through complementary feeding.

The onset of weaning is influenced by several factors that contribute to the infant's autonomy, such as proper neuromotor development, development of taste and personal inclinations, maturation of kidney and gastrointestinal function, and social and socioeconomic factors.1 This gradual process can last from a few months to a couple of years.

There are different types of weaning, which vary according to traditions, ethnicity and scientific currents. These include traditional weaning or TSF, Baby-led Weaning (BLW) and Baby-led introduction to solids (BLISS).

TSF consists of the introduction of complementary feeding including solid or semisolid type foods served in the form of spoon puree and specially prepared foods for children with suggested doses, composition, quantities, and schedules.

BLW or autodiving refers to a type of complementary feeding introduction in which the infant can control the process from the beginning, setting the pace according to his or her appetite. The introduction of food is dictated by the infant's interest in food and his or her ability to self-feed small portions of food normally taken during family meals. For this purpose, the infant sits at the table with family members and takes food portions of a size and texture proportionate to his or her neurodevelopment and acquisition. The infant may feed independently with or without the aid of cutlery.

BLISS is a modified form of BLW that has implemented arrangements aimed at preventing foreign body inhalation. This modified version includes the start of weaning at the age of 6 months, coupled with general advice and rules specifically created to reduce the risk of choking. Pediatricians of free choice (PLS) play a key role in the implementation of weaning, in terms of providing advice on the different modes and food selection and preparation.

Benefits and risks related to different types of weaning BLW reduces the risk of eating disorders, facilitates the transition to the family diet, and incentivizes the family to follow a balanced diet.

This practice promotes the infant's adaptation to different food textures and tastes, speeds up learning to chew, development of fine motor skills, and overall maturation of the child, and is not correlated with poor infant staturo-ponderal growth. Although this approach has many advantages, a theoretical concern, relates to its safety and the possible increased risk of choking and inhalation from EC. There are conflicting data in the literature; some studies point to a likely reduction in the risk of choking due to an increase in gagging, which would lead to regurgitation of food rather than inhalation of food. In fact, BLW is an approach in which the infant tends to assume a more appropriate posture and is focused on actively chewing foods, unlike traditional weaning in which he or she receives, in a more relaxed position, foods served in pureed form that are directly swallowed without being chewed. So, according to some authors, traditional weaning would stimulate the infant's chewing ability less and increase the risk of inhalation compared with BLW. According to other authors, children following a BLISS-type weaning method accompanied by advice to minimize choking risks do not have a higher risk of inhalation than children following traditional weaning. This would show that the safety of TSF and BLISS may be comparable. In light of these observations, it is of particular interest to investigate this topic further given the absence of sufficient evidence in the literature that has clarified the relationship between these issues and weaning patterns.

ELIGIBILITY:
Inclusion Criteria:

Parents group:

* Overage parents with children between the ages of 4 and 18 months
* Need to have an electronic tool that allows direct access to the link connected to an internet network
* Understanding of the Italian language
* Obtaining informed consent from the parent completing the questionnaire

Pediatricians group:

* Activities of Free Choice Pediatrician in Italy.
* Need to have an electronic tool that allows direct access to the link connected to an Internet network
* Obtaining informed consent

Exclusion Criteria:

Parents group:

- Parents of children with chronic neurological diseases, dysphagia, chronic diseases involving specific diet, intestinal diseases resulting in malabsorption;

Pediatricians group:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participation will be offered to all parents who reflect the inclusion criteria by specifying the observational nature of the study and the importance of deepening the prevalence and knowledge of the different diveating modes. It is specified that one of the two parents will be sufficient to complete the questionnaire. In the case of twins, the questionnaire will include completion of the weaning questions for each child. These persons will be recruited from the wards and waiting rooms of the Centers participating in the study without retaining any personal data of the enrolled subject. Access to the online questionnaire will be via access link that will be provided to the subjects via e-mail to the address they provide.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate how parents and pediatricians implement weaning | through study completion, an average of 1 year
  * Percentage of parents choosing a particular weaning mode;
  * reasons expressed by Pediatricians of Free Choice in suggesting their chosen weaning mode.

SECONDARY OUTCOMES:
Different ways of weaning suggestionated by free choice Pediatricians | through study completion, an average of 1 year
  * Analysis of the different ways in which weaning is implemented in terms of food choice and meal delivery by parents and related suggestions by Free Choice Pediatricians;
  * What risks associated with weaning are perceived by parents and Pediatricians of Free Choice.

CONTACTS AND LOCATIONS:
Overall Officials: Arianna Dondi, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (4):
- Italy (4):
  - Ospedale S. Maria della Scaletta, Azienda USL di Imola UO Pediatria, Imola, Bologna
  - Ospedale Ramazzini di Carpi, Azienda USL di Modena UO Pediatria, Carpi, Modena
  - Ospedale Maggiore, Azienda USL di Bologna UO Pediatria, Bologna
  - IRCCS Azienda Ospedaliero - Universitaria di Bologna, U.O. Pediatria d'Urgenza, Pronto Soccorso e Osservazione Breve ed Intensiva, Bologna